CLINICAL TRIAL: NCT03220984
Title: Open-label, Single Center, Phase Ⅱ Clinical Trial to Evaluate Safety and Efficacy of Immuncell-LC in the Patients for Refractory Metastatic Colorectal Cancer
Brief Title: The Safety and Efficacy Test of Immuncell-LC to Treat Refractory Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Seung Hyuk Baik, Principal Investigator, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2016-0346
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy group (Experimental): All enrolled patients receive a total of 12 times of Immuncell-LC therapy
  Interventions: Biological: Immuncell-LC intravenous infusion using a CIK cell agent

INTERVENTIONS:
Biological: Immuncell-LC intravenous infusion using a CIK cell agent — Patients with metastatic colorectal cancer, which is refractory to the 3rd-line chemotherapy are enrolled in this study. Enrolled patients receive a total of 12 times of Immuncell-LC therapy: 8 times in every 1 week and the next 4 times in every 2 weeks. The treatment responses of immuncell-LC are evaluated by radiologic findings (Abdomin-pelvic CT and Chest CT), immune-markers and a selorogic tumor marker (Carcinoembryologic antigen (CEA)) at the 8th week and 17th week. The safety of Immuncell-LC is evaluated by the results of serologic tests, vital signs, ECOG-PS and adverse events. The follow-up period is the 1 year after the enrolled date.

SUMMARY:
This study aims to evaluate the safety and efficacy of Immuncell-LC, the adoptive immuntherapeutic agent composed of a CIK cell agent, to treat patients with metastatic colorectal cancer, which are refractory to the 3rd-line chemotherapeutic agents.

All enrolled patients received the 12 times of Immuncell-LC therapy: 8 times in every 1 week and 4 times in every 2 weeks.

DETAILED DESCRIPTION:
Stage IV colorectal cancer(CRC) has poor survival rate in spite of the development of chemotherapeutic agents. It is regarded as a standard palliative chemotherapy using with both targeted agents and cytototic chemotherpeutic agents. However, it is still demanding to treat stage IV CRC patients, who are refractory responses in these chemotherapeutics. In addition, patients were suffered from the various adverse events by the repetive cytotoxic chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years old
* Clinical diagnosis of metastatic colon cancer or rectal cancer
* ECOG ≥ 2
* ASA ≤ 3
* Patients should meet below conditions by serologic test, kidney and liver function test: Re-evaluation is permitted during screening.

  * Absolute neutrophil count (ANC) ≥ 1500/μL
  * Hemoglobin level ≥ 9.0 g/dL
  * Platelet count >75,000/μL
  * BUN and serum Creatinine are less than or equal to 1.5 multiply normal upper-limit
  * AST and ALT are less than 2.5 multiply normal upper-limit (If a patients has liver metastases, AST and ALT are less than 5 times of normal upper-limits.)

Exclusion Criteria:

* Patient who has disease history of immune deficiency or auto-immune disease (ex. Multiple sclerosis, arthritis rheumatism, Buerger's disease, and adolescent-occurred insulin dependent diabetes)
* Pateint who diagnosed immune-deficiency diseases
* Diagnosis of malignant tumor within 5 years before this clinical trial. (except for skin cancer, local prostate canter or carcinoma in situ of the cervix
* Patient who needs interventional therapy due to intestinal obstruction of obstructive jaundice
* Diagnosed status of infection or sepsis
* Uncontrolled hypertension or heart-failure
* Severe allergic history, which is diagnosed by sub-investigators
* Serious psychologic disease, which is diagnosed by sub-investigators
* Pregnant women, nursing mother or people who has intention of being preganant during the clinical test
* Patient who participated in other clinical trials within last 4 weeks before this trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
the disease control rate (DCR) | 4 months (17 weeks)
  To evaluate the disease control rate (DCR) : complete reponse(CR), partial response(PR), stable disease(SD).

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyuk Baik, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea